CLINICAL TRIAL: NCT00188435
Title: A Comparison of Chest Radiography and Minimum Dose Chest CT
Brief Title: Comparison of CXR and MnDCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0731
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2005-09

CONDITIONS: Acute Dyspnoea

INTERVENTIONS:
Procedure: Minimum Dose CT

SUMMARY:
A comparison of chest x-ray (CXR) and Minimum dose CT (MnDCT) in the acutely ill patient. The hypothesis is that MnDCT is more sensitive than CXR in the detection of acute findings in the acutely ill patient.

DETAILED DESCRIPTION:
A comparison of chest x-ray (CXR) and Minimum dose CT (MnDCT) in a cohort of 100 patients admitted for acute respiratory distress. Chest radiography (CXR) is compared to Minimum Dose CT (MnDCT) for the detection of consolidation;lung nodules, heart failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for investigation of acute pulmonary embolus

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-11; Study Completion 2004-12

PRIMARY OUTCOMES:
A comparison of CXr and MnDCT in the detection of acute findings within the thorax

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto